CLINICAL TRIAL: NCT02281929
Title: Evaluation of the Efficacy of an Antibiotic Combined With Standard Treatment in Severe Alcoholic Hepatitis
Brief Title: Efficacy of Antibiotic Therapy in Severe Alcoholic Hepatitis Treated With Prednisolone
Acronym: AntibioCor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014_05; 2014-002536-13 (EudraCT Number); PHRC-2013-0552 (Other: Minister of Health, France)
Record Dates: First submitted 2014-10-28; First posted 2014-11-04 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2021-03

CONDITIONS: Alcoholic Hepatitis; Alcoholic Liver Disease
Keywords: Alcoholic hepatitis; corticotherapy; antibiotherapy; survival; infection; hepato renal syndrome
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Diseases, Alcoholic; Infections; Hepatorenal Syndrome | interventions — Amoxicillin; Amoxicillin-Potassium Clavulanate Combination; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- amoxicillin+ prednisolone (Active Comparator): Oral antibiotherapy during 30 days using amoxicillin+clavulanic acid at a daily dose of 3 gram (amoxicillin) and 375 mg (clavulanic acid) in three daily doses of 1g/125mg. Oral corticotherapy during 30 days with prednisolone at 40 mg/j in a single daily dose in the morning.
  Interventions: Drug: Amoxicillin; Drug: Prednisolone
- Placebo + prednisolone (Placebo Comparator): Oral placebo of amoxicillin- clavulanic acid in three daily doses during 30 days Oral corticotherapy during 30 days with prednisolone at 40 mg/j in a single daily dose in the morning.
  Interventions: Drug: Placebo; Drug: Prednisolone

INTERVENTIONS:
Drug: Amoxicillin — Amoxicillin+clavulanic acid at a daily dose of 3 gram / 375 mg in three daily doses of 1g/125mg, during 30 days
  Other Names: Amoxicillin + clavulanic acid
  Arms: amoxicillin+ prednisolone
Drug: Placebo — Placebo in three daily doses during 30 days
  Other Names: Placebo of amoxicillin
  Arms: Placebo + prednisolone
Drug: Prednisolone — Prednisolone at 40 mg/j in a single daily dose in the morning, during 30 days
  Other Names: corticotherapy

SUMMARY:
Treatment of reference of severe alcoholic hepatitis is based on corticosteroids, given for 28 days. However, about 25-35% of patients do not take benefit from this treatment and die within the 6 months following the diagnosis. Numerous trials have evaluated the impact of several strategies in association with corticosteroids. None of them has shown an improvement in survival (primary endpoint) as compared to corticosteroids alone.

The project is based on an approach never tested in a randomized controlled trial in severe alcoholic hepatitis, targeting the group of patients at high risk of death (25-35% at 2 months). This approach is based on animal and human studies.Antibiotics are effective in animal models and in other circumstances characterized by liver failure such as gastrointestinal bleeding related to portal hypertension. The interest of studying this population is emphasized by the frequency of infections in these critically ill patients. Antibiotics will be administered before the development of any infection, as it is likely that these patients present with mesenteric bacterial adenitis without systemic signs of infection. Primary endpoint will be 2-month survival as most deaths occur within 60 days and treatment is given for 30 days.

DETAILED DESCRIPTION:
This is a multicenter double-blind randomized controlled study on two parallel groups.

Once inclusion and exclusion criteria verified and after having obtained patient written consent, participative centers will process to inclusion in the trial.

Corticosteroids as well as antibiotics or their placebo will be started orally. Patients will be managed in the hospital unit until day 7, which corresponds to the evaluation of response to treatment using the Lille model. After this 7-day period, patients will be followed-up at day 14, day 21, day 30, day 60 (primary endpoint).

During each visit, biological and clinical features including efficacy and tolerance will be assessed as well as presence of infection and hepatorenal syndrome (secondary endpoints).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75
* Recent onset of jaundice (<3 months)
* Biopsy proven alcoholic hepatitis (transjugular liver biopsy)
* Maddrey's discriminant function ≥ 32, defining severe alcoholic hepatitis
* MELD score ≥21
* Alcohol consumption ≥ 40g/day (women) and ≥ 50g/day (men)
* Written informed consent

Exclusion Criteria:

* Previous severe allergy or hypersensitivity to amoxicillin or clavulanic acid (anaphylactic shock, Quincke edema, severe urticaria)
* Hypersensitivity to any component of the medication
* History of liver injury to amoxicillin and/or clavulanic acid
* Phenylketonuria, because of the presence of aspartame in the powder for the oral suspension
* Type 1 hepatorenal syndrome before the initiation of treatment
* Severe extrahepatic disease
* Any malignant tumor < 2 years
* Uncontrolled gastrointestinal bleeding
* Ongoing viral or parasitic infection
* Untreated bacterial infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2015-06-13 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Patient alive | at day 60
  The percentage of patients alive at 2 months in the experimental arm compared to the percentage of patients alive in the control arm

SECONDARY OUTCOMES:
Infection | at day 7, day14, day 21, day 30, day 60; at 3 months, at 6 months
  incidence of infection over the 2-month period in the antibiotic+corticosteroid arm as compared to the control arm
Hepatorenal syndrome | at day 7, day14, day 21, day 30,at 3 months, at 6 months
  incidence of hepatorenal syndrome over the 2-month period in the antibiotic+corticosteroid arm as compared to the control arm
MELD score <17 | at day 7, day14, day 21, day 30,
  percentage of patients with a low risk of mortality during the first two months (assessed by a MELD score <17) in the two arms of treatment. The MELD score will be calculated using the following formula:(9.57 × log creatinine in milligrams per deciliter) + (3.78 × log bilirubin in milligrams per deciliter) + (11.20 × log international normalized ratio) + 6.43.
Lille Model | at day 7, after the first administration of treatment
  percentage of patients disclosing a response to treatment assessed by the Lille model (<0.45) in the two arms of treatment.
Patient alive | at 3 months, at 6 months
  The percentage of patients alive at 2 months in the experimental arm compared to the percentage of patients alive in the control arm

CONTACTS AND LOCATIONS:
Overall Officials: Mathurin Philippe, MD,PhD, Study Chair — University Hospital, Lille
Locations (20):
- France (20):
  - CHU d'Amiens, Amiens
  - CHU, Angers
  - CHU de Besançon, Besançon
  - Hôpital Jean Verdier (AH-HP), Bondy
  - CHU de Caen, Caen
  - Hôpital BEaujon (AP-HP), Clichy
  - Centre hospitalier, Dunkirk
  - CHU Grenoble, Grenoble
  - Hôpital Claude Huriez, CHU, Lille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Hôpital Saint Antoine (AP-HP), Paris
  - Hôpital La Pitié (AP-HP), Paris
  - CHU Poitiers, Poitiers
  - CHU Pontchaillou, Rennes
  - CHU, Rouen
  - CHU, Toulouse
  - Centre Hospitalier, Valenciennes
  - Hôpital Paul Brousse (AH-HP), Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathurin P, O'Grady J, Carithers RL, Phillips M, Louvet A, Mendenhall CL, Ramond MJ, Naveau S, Maddrey WC, Morgan TR. Corticosteroids improve short-term survival in patients with severe alcoholic hepatitis: meta-analysis of individual patient data. Gut. 2011 Feb;60(2):255-60. doi: 10.1136/gut.2010.224097. Epub 2010 Oct 12. PMID 20940288
- [Background] Nguyen-Khac E, Thevenot T, Piquet MA, Benferhat S, Goria O, Chatelain D, Tramier B, Dewaele F, Ghrib S, Rudler M, Carbonell N, Tossou H, Bental A, Bernard-Chabert B, Dupas JL; AAH-NAC Study Group. Glucocorticoids plus N-acetylcysteine in severe alcoholic hepatitis. N Engl J Med. 2011 Nov 10;365(19):1781-9. doi: 10.1056/NEJMoa1101214. PMID 22070475
- [Background] Lucey MR, Mathurin P, Morgan TR. Alcoholic hepatitis. N Engl J Med. 2009 Jun 25;360(26):2758-69. doi: 10.1056/NEJMra0805786. No abstract available. PMID 19553649
- [Background] Louvet A, Wartel F, Castel H, Dharancy S, Hollebecque A, Canva-Delcambre V, Deltenre P, Mathurin P. Infection in patients with severe alcoholic hepatitis treated with steroids: early response to therapy is the key factor. Gastroenterology. 2009 Aug;137(2):541-8. doi: 10.1053/j.gastro.2009.04.062. Epub 2009 May 13. PMID 19445945
- [Background] Louvet A, Naveau S, Abdelnour M, Ramond MJ, Diaz E, Fartoux L, Dharancy S, Texier F, Hollebecque A, Serfaty L, Boleslawski E, Deltenre P, Canva V, Pruvot FR, Mathurin P. The Lille model: a new tool for therapeutic strategy in patients with severe alcoholic hepatitis treated with steroids. Hepatology. 2007 Jun;45(6):1348-54. doi: 10.1002/hep.21607. PMID 17518367
- [Background] Mathurin P, Louvet A, Duhamel A, Nahon P, Carbonell N, Boursier J, Anty R, Diaz E, Thabut D, Moirand R, Lebrec D, Moreno C, Talbodec N, Paupard T, Naveau S, Silvain C, Pageaux GP, Sobesky R, Canva-Delcambre V, Dharancy S, Salleron J, Dao T. Prednisolone with vs without pentoxifylline and survival of patients with severe alcoholic hepatitis: a randomized clinical trial. JAMA. 2013 Sep 11;310(10):1033-41. doi: 10.1001/jama.2013.276300. PMID 24026598
- [Result] Louvet A, Labreuche J, Dao T, Thevenot T, Oberti F, Bureau C, Paupard T, Nguyen-Khac E, Minello A, Bernard-Chabert B, Anty R, Wartel F, Carbonell N, Pageaux GP, Hilleret MN, Moirand R, Nahon P, Potey C, Duhamel A, Mathurin P. Effect of Prophylactic Antibiotics on Mortality in Severe Alcohol-Related Hepatitis: A Randomized Clinical Trial. JAMA. 2023 May 9;329(18):1558-1566. doi: 10.1001/jama.2023.4902. PMID 37159035
- See also: Related Info — http://www.lillemodel.com/